CLINICAL TRIAL: NCT00398970
Title: Diagnostic Utility of Endobronchial Ultrasound in the Investigation of Suspected Malignant Lung Lesions Where the Lesions Are Not Visible During Bronchoscopy.
Brief Title: Utility of Endobronchial Ultrasound in the Investigation of Suspected Lung Cancer.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: Helse Sunnmore, 6026 Ålesund (Unknown)
Responsible Party: Jon Andrew Hardie, MD/PhD, Haukeland Univiersity Hospital, Bergen, Norway
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 12562
Record Dates: First submitted 2006-11-13; First posted 2006-11-14 (Estimated); Last update posted 2008-02-29 (Estimated); Status verified 2008-02

CONDITIONS: Lung Cancer
Keywords: Endobronchial ultrasonography; Fluoroscopy; Guide sheath; Peripheral pulmonary lesion; Transbronchial biopsy
MeSH Terms: conditions — Lung Neoplasms

ARMS (2):
- Traditional flouroscopy guided sampling (Active Comparator)
  Interventions: Device: Endobronchial ultrasound miniprobe
- Ultrasound guide sampling (Experimental)
  Interventions: Device: Endobronchial ultrasound miniprobe

INTERVENTIONS:
Device: Endobronchial ultrasound miniprobe — Endobronchial ultrasound miniprobe is used to identify solid mass in lung parenchyma.

SUMMARY:
Bronchoscopy of non visible lesions in the lung, have a low diagnostic yield. The use of endoscopic ultrasound might increase the diagnostic yield. This prospective study randomises between bronchoscopy with the use of a ultrasound miniprobe and bronchoscopy without the use of a miniprobe in clinical practice at Haukeland University Hospital.

The study hypothesis:

The use of the ultrasound miniprobe will increase the diagnostic yield of bronchoscopy in non visible lesions.

DETAILED DESCRIPTION:
Bronchoscopy is usually the primary investigation of lesions in the lung. X-ray fluorescence guides the sampling with brushing, biopsy or trans bronchial needle aspiration (TBNA) if the lesion not is visible. Ct guided trans-thoracic sampling will be performed if a the sample is non representative. This will delay the diagnosis, and trans-thoracic sampling has a higher risk of pneumothorax. The use of a ultrasound miniprobe might increase the diagnostic yield of bronchoscopy in non visible lesions. The ultrasound probe in a guide sheath is advanced to the lesion with use of X-ray fluorescence. When the lesion is visualised the miniprobe is removed and sampling is performed with TBNA, biopsy and brushing through the guide sheath. If rapid on site cytoevaluation is negative, new TBNA is performed. Previous trials have shown a diagnostic yield without ultrasound between 40-50% and with ultrasound between 60-80%. The studies with ultrasound have been performed by "super specialists". This study will evaluate bronchoscopy with the use of ultrasound miniprobe in clinical practice without "super specialists". It is a prospective randomised trial.

ELIGIBILITY:
Inclusion Criteria:

* All patients with lesions suspicious of malignancy in the lung.

Exclusion Criteria:

* Patients with lesions assumed to be visible by bronchoscopy.
* Later proven visible lesion by bronchoscopy.
* Patients not able to be investigated by bronchoscopy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2005-06; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield of bronchoscopy | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jon A Hardie, MD/PhD, Principal Investigator — Department of Thoracic Medicine, Haukeland University Hospital
Locations (1):
- Department of Thoracic Medicine, Bergen, Norway

REFERENCES:
- [Background] Kikuchi E, Yamazaki K, Sukoh N, Kikuchi J, Asahina H, Imura M, Onodera Y, Kurimoto N, Kinoshita I, Nishimura M. Endobronchial ultrasonography with guide-sheath for peripheral pulmonary lesions. Eur Respir J. 2004 Oct;24(4):533-7. doi: 10.1183/09031936.04.00138603. PMID 15459129
- [Background] Kurimoto N, Miyazawa T, Okimasa S, Maeda A, Oiwa H, Miyazu Y, Murayama M. Endobronchial ultrasonography using a guide sheath increases the ability to diagnose peripheral pulmonary lesions endoscopically. Chest. 2004 Sep;126(3):959-65. doi: 10.1378/chest.126.3.959. PMID 15364779
- [Background] Herth FJ, Ernst A, Becker HD. Endobronchial ultrasound-guided transbronchial lung biopsy in solitary pulmonary nodules and peripheral lesions. Eur Respir J. 2002 Oct;20(4):972-4. doi: 10.1183/09031936.02.00032001. PMID 12412691
- [Background] Schreiber G, McCrory DC. Performance characteristics of different modalities for diagnosis of suspected lung cancer: summary of published evidence. Chest. 2003 Jan;123(1 Suppl):115S-128S. doi: 10.1378/chest.123.1_suppl.115s. PMID 12527571
- [Background] Baaklini WA, Reinoso MA, Gorin AB, Sharafkaneh A, Manian P. Diagnostic yield of fiberoptic bronchoscopy in evaluating solitary pulmonary nodules. Chest. 2000 Apr;117(4):1049-54. doi: 10.1378/chest.117.4.1049. PMID 10767238